CLINICAL TRIAL: NCT01953250
Title: To Assess the Functional Outcome in Patients That Underwent Laparoscopic Sigmoid and/or Rectum Resection
Brief Title: Functional Outcome in Patients That Underwent Laparoscopic Sigmoid and/or Rectum Resection
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S-54351
Record Dates: First submitted 2013-02-19; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2012-04

CONDITIONS: Endometriosis
Keywords: Deep infiltrating endometriosis; Laparoscopic sigmoid resection; laparoscopic rectum resection; Colorectal surgery
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infiltrating endometriosis: 272 patients that underwent laparoscopic sigmoid and/or rectum resection with the indication of deep infiltrating endometriosis, in the department of Abdominal Surgery, University Hospital Leuven, between the year 1997 and September 2011.

SUMMARY:
Questionnaire To assess the functional outcome in patients that underwent laparoscopic sigmoid and/or rectum resection.

DETAILED DESCRIPTION:
A questionnaire will be sent to every patient by mail. The questionnaire that will be used is the COREFO questionnaire (ColoRectal Functional Outcome).

Depending on the amount of responses, we will try to make connections between peri-operative data and functional outcome after considerable period of follow-up. Peri-operative factors include grade of endometriosis, surgical technique and post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent laparoscopic sigmoid and/or rectum resection with the indication of deep infiltrating endometriosis

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 272 patients that underwent laparoscopic sigmoid and/or rectum resection with the indication of deep infiltrating endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
ColoRectal Functional Outcome | 1 day
  Operation: between 1997 and 2011 Questionnaire to assess the colorectal function sent once in 2012

CONTACTS AND LOCATIONS:
Overall Officials: André JL D'Hoore, PhD, Principal Investigator — University Clinics Gasthuisberg Department of Abdominal Surgery
Locations (1):
- University Clinics Gasthuisberg, Leuven, Flemish Brabant, Belgium